CLINICAL TRIAL: NCT02286882
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Single Ascending Oral Doses Of Pf-06409577 In Healthy Adult Subjects
Brief Title: A Single Oral Dose Study Of PF-06409577 In Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated prematurely on June 19, 2015 for business reasons. There were no safety concerns in the study which led to the decision.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7881001; FIH (Other: Alias Study Number); 2014-004022-18 (EudraCT Number)
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Single Ascending Dose; healthy subjects
MeSH Terms: interventions — PF-6409577

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 2: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 3: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 4: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 5: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 6: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 7: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 8: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo
- Cohort 9: PF-06409577 or placebo (Experimental): Single ascending doses of PF-06409577 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06409577 or Placebo

INTERVENTIONS:
Drug: PF-06409577 or Placebo — PF-06409577or placebo will be administered as an extemporaneously prepared suspension once in each cohort

SUMMARY:
PF-06409577 is a new compound proposed for the treatment of diabetic nephropathy. The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single oral doses of PF-06409577 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 18 to 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

- Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | 0-48 hours post dose
Number of Participants With Laboratory Test Values of Potential Clinical Importance | 0-48 hours post dose
Number of Participants With Vital Signs Findings (Including Bood Pressure and Pulse Rate) of Potential Clinical Importance | 0-48 hours post dose
Number of Participants With Electrocardiogram (ECG) Findings of Potential Clinical Importance | 0-48 hours post dose
Number of Participants With Echocardiogram Findings of Potential Clinical Importance | 0-48 hours post dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Time 24 hours (AUC24) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post dose
  Area under the plasma concentration time-curve from zero to time 24 hours post dose (AUC24)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - infinity)] for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  AUC (0 - infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Maximum Observed Plasma Concentration (Cmax) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Apparent Oral Clearance (CL/F) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06409577 | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Total amount of PF-06409577 excreted in the urine over 24 hours (Ae24) | 0-24 hours post dose
  Total amount of unchanged drug excreted in the urine over 24 hours.
Total amount of PF-06409577 excreted in the urine over 24 hours, expressed as percent of dose (%Ae24) | 0-24 hours post dose
  Total amount of unchanged drug excreted in the urine over 24 hours, expressed as percent of dose.
Renal clearance for PF-06409577 | 0-24 hours post dose
  Renal clearance of a drug is a measure of the rate at which a drug is excreted unchanged into urine.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium